CLINICAL TRIAL: NCT01378845
Title: Monocenter, IIT, Open Controlled and Prospectiv Study to Define the Prognostic Influence of Light Rheography Measurement of Patients With Secundary Raynaud Syndrome With Ulcers at Fingertips Throughout the Medicinal Therapy
Brief Title: Prognostic Influence of Light Rheography Measurement of Patients With Secondary Raynaud Syndrome With Ulcers on Hands
Acronym: Anti-Vasospasm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christoph Hehrlein (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor-Investigator, Christoph Hehrlein, Professor Dr. med., University of Freiburg
Organization: University of Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-002127-17
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Raynaud's Phenomenon; Skin Necrosis
Keywords: Morbus Raynaud; Ulcera Hands, Toes; Vasospastic disorder; Raynaud's phenomenon
MeSH Terms: conditions — Raynaud Disease; Necrosis | interventions — Bosentan; Alprostadil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prostavasin (Placebo Comparator)
  Interventions: Drug: Prostavasin
- Prostavasin + Bosentan (Active Comparator)
  Interventions: Drug: Tracleer; Drug: Prostavasin

INTERVENTIONS:
Drug: Tracleer — 14 days 62,5 mg Bosentan p.o 140 days 125 mg Bosentan p.o
  Other Names: Bosentan
  Arms: Prostavasin + Bosentan
Drug: Prostavasin — Prostavasin 60 µg i.v, 5 days per week for 2 weeks
  Other Names: Aprostadil

SUMMARY:
The purpose of this study is to evaluate the prognostic influence of light rheography measurement at the fingertips from subjects with secundary Raynaud syndrome.

DETAILED DESCRIPTION:
Digital Ulcers (DU) belong to one of the most prevalent complications of systemic scleroses, leading in course to considerable impairment in everyday and professional life. The aetiology of the emergence of DU in patients with systemic scleroses (SSc) is complex, whereas the disease itself is primarily characterized by a vasculopathy of the small arterial vessels. In the course of the disease this chronic infection leads to fibrotic intimal hyperplasia, adventitial fibrosis, and thus to a significant lumen narrowing. So far, a number of independent risk factors have been identified, such as male gender, chronic infections of the esophagus, pulmonary-arterial hypertension, evidence of specific antibodies (e.g. anti-Scl70) in the blood, or the a previous manifestation of a Raynoud Syndrom.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Limited or diffuse systemic sclerosis/scleroderma with at least one ulcera at fingertip
* Age > 18 Years
* Weight > 40 Kg

Exclusion Criteria:

* Sympathectomy
* Ulcers due to other condition (PVD, DM, Thromboangiitis obliterans etc.)
* Antibiotic concomitant medication
* Therapy with Prostanoids within the last 4 weeks
* Previous Bosentan therapy
* Severe liver and renal insufficiency(creatinin >2.0 mg/dl;AST/ALT > 3X UNL)
* severe cardiac- pulmonal diseases
* Untreated or therapy refractory Hypertension
* Noncompliance
* Pregnancy or nursing (Pregnancy test required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Quantification of the blood flow before, during and after the medical therapy | 24 weeks
  The primary objective of this study is defined by the dynamics of the (post)capillary blood flow before (baseline value) and 12 weeks after treatment, measured by means of the LRR. In doing so, the therapeutic effect, in terms of the change in (post)capillary blood flow after treatment compared to baseline value, is to be quantitatively determined.

SECONDARY OUTCOMES:
Emerge of new ulcers | > 24 weeks
  Additionally, it is to be examined if new DUs emerge after 24 weeks or not. The prospects for recovery of the DU will be investigated by means of visual analogue scale (VAS), photo-documentation, and D-LRR after 2, 6, 12, and 24 weeks of medicinal therapy. Furthermore, as mentioned above, the change in the HIF-1alpha gene expression before (baseline value) and 6 weeks after treatment is to be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kerber, Dr. med., Principal Investigator — Universitätsklinik Freiburg
Locations (1):
- University Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] -Distler O, Gay S. [Scleroderma]. Internist (Berl) 2010; 51(1):30-38. -Mouthon L, Mestre-Stanislas C, Berezne A et al. Impact of digital ulcers on disability and health-related quality of life in systemic sclerosis. Ann Rheum Dis 2010; 69(1):214-217. -Denton C, Krieg T, Guillevin L. The burden of complications in patients with digital ulcers (DU) and systemic sclerosis (SSc): Preliminary findings from the DUO-Registry. 2009: 273. -Korn JH, Mayes M, Matucci CM et al. Digital ulcers in systemic sclerosis: prevention by treatment with bosentan, an oral endothelin receptor antagonist. Arthritis Rheum 2004; 50(12):3985-3993. -Block JA, Sequeira W. Raynaud's phenomenon. Lancet 2001; 357(9273):2042-2048.
- [Background] -Sunderkotter C, Herrgott I, Bruckner C et al. Comparison of patients with and without digital ulcers in systemic sclerosis: detection of possible risk factors. Br J Dermatol 2009; 160(4):835-843. -Muller-Ladner U. Akrale Ischämiesyndrome: vom Raynaud-Syndrom zur systemischen Sklerose. Bremen/London/Boston: UNI-MED Verlag AG, 2009 -Arab A, Kuemmerer K, Wang J et al. Oxygenated perfluorochemicals improve cell survival during reoxygenation by pacifying mitochondrial activity. J Pharmacol Exp Ther 2008; 325(2):417-424. -Pope J, Fenlon D, Thompson A et al. Iloprost and cisaprost for Raynaud's phenomenon in progressive systemic sclerosis. Cochrane Database Syst Rev 2000;(2):CD000953. -Kawald A, Burmester GR, Huscher D et al. Low versus high-dose iloprost therapy over 21 days in patients with secondary Raynaud's phenomenon and systemic sclerosis: a randomized, open, single-center study. J Rheumatol 2008; 35(9):1830-1837. -Kowal-Bielecka O, Landewe R, Avouac J et al. EULAR recommendations for the treatment of systemic sclerosis: a report from the EULAR Scleroderma Trials and Research group (EUSTAR). Ann Rheum Dis 2009; 68(5):620-628. -Sunderkotter C, Riemekasten G. [Raynaud phenomenon in dermatology:Part 2:therapy]. Hautarzt 2006; 57(10):927-938. -Ludwig M. Angiologie in Klinik und Praxis. 1 ed. Stuttgart: Thieme Verlag, 1998; 1-334.